CLINICAL TRIAL: NCT02983409
Title: A Study of Analysis the Relationship Between the Findings of Abdominal Comptuted Tomography and the Clinical Outcomes in Acute Urinary Stone Patients
Brief Title: Analysis the Relationship Between the Abdomen CT and Outcomes in Acute Urinary Stone Patients
Status: Completed | Type: Observational
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Sang O, Park, Assistant Professor, Konkuk University Medical Center
Other Study IDs: UstoneCT
Record Dates: First submitted 2016-10-26; First posted 2016-12-06 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Urinary Calculi; Emergency Service, Hospital
Keywords: computerized tomography; Urinary Calculi; Patient admission; Pain
MeSH Terms: conditions — Urinary Calculi; Emergencies; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pstone: Adult Patients (> 18years) who were diagnosed as the urinary stone in the ED. All patients who visited the ED with compalin of acute pain, and urinary stone was idenfied by urinary CT in the ED.
  Interventions: Radiation: Pstone

INTERVENTIONS:
Radiation: Pstone — A adult patients who were diagnosed as urinary stone by the urinary CT

SUMMARY:
This is an observational study based on retrospectively collected data of ureter stone patients between 2011 and 2014. Aim of study is to determine radiologic findings of non-contrast abdominal computerized tomography as predicting clinical outcomes of suspect ureter stone patients in emergency department (ED).

DETAILED DESCRIPTION:
Gennerally, non-contrast abdominal computerized tomography is a choice of diagnosis for a ureter stone patient.There was no known well of efficacy of CT for predicting the outcomes in ureter stone patient in ED.

Hypothesis of this study are some findings of non-contrast CT may be helpful to predict the clinical outcomes of pain severity (multidose of painkiller), admission and revisit to ED within 5 days after discharge. Investigators analyzed multiple variables including age, sex, initial clinical findings, and various CT findings to assess their association with outcomes; multidose of painkiller in ED, admission at ED and revisit to ED within 5 days.

ELIGIBILITY:
Inclusion Criteria:

* ED Patients
* Age > 18 years
* Confirmed the ureter stone by Abdomen or Urinary CT

Exclusion Criteria:

* Known a uninary congenital or acquired anomaly
* combined other healthy preblem at the ED

  * infection, renal dysfunction et al
* Known the chronic disease : Hypertension ,Diabetes, Tuberculosis, Malignance et al

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A adult (>18 years) patients who was diagnosed as ureter stone. They had no previous history of ureter stone within recent 1 year. They should not have a uninary congenital or acquired anomaly and chronic renal disease.
Sampling Method: Non-Probability Sample
Enrollment: 862 (Actual)
Dates: Start 2011-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Multiple-painkiller | within 6 hours after the ED visit
  Patient who take the over 2 painkiller medication because of serious pain.
Admission at ED | within 24 hours after the ED visit
  Patient who admitted at the ED
Revisit to the hospital within 5 days | within 5 days after the ED discharge
  Patient who revisit the hospital within 5 days after the ED discharge

CONTACTS AND LOCATIONS:
Overall Officials: Sang O Park, Dr, Principal Investigator — 1Department of Emergency Medicine, School of Medicine, Konkuk University, Konkuk University Medical Center

IPD SHARING:
Plan to Share IPD: No